CLINICAL TRIAL: NCT00900666
Title: Randomized Controlled Trial on the Effects of Botulinum Toxin Injections in the Rectus Femoris on Gait Function in Stiff Knee Gait Following Acquired Brain Injury
Brief Title: Efficacy of Botulinum Toxin Injections in the Rectus Femoris to Treat Stiff Knee Gait Following Acquired Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original subject recruitment goal was unrealistic. Study was terminated at N=19.
Sponsor: Mary Free Bed Rehabilitation Hospital (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Krisanne B. Chapin, PhD, Manager and Clinical Biomechanist, Mary Free Bed Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFB2008.08
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Stiff Knee Gait; Brain Injuries
Keywords: Stiff knee gait; Gait analysis; Traumatic Brain Injury; Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline injection (Placebo Comparator)
  Interventions: Drug: placebo
- Botulinum toxin injection (Experimental)
  Interventions: Drug: botulinum toxin A (BTX-A)

INTERVENTIONS:
Drug: placebo — A total of 2 cc sterile normal saline: will be injected in 0.5 cc aliquots into 4 different injectate sites within the rectus femoris (with EMG guidance) of the involved limb.
  Arms: Saline injection
Drug: botulinum toxin A (BTX-A) — 200 Units BTX-A reconstituted with 2 cc sterile normal saline in 100:1 ratio. Teflon-coated EMG guidance for confirmation of injection into the Rectus femoris muscle in addition to utilizing standardized injection landmarks, the solution will be injected in 0.5 cc aliquots into 4 different injectate sites within the muscle.
  Arms: Botulinum toxin injection

SUMMARY:
Stiff knee gait is a common gait dysfunction following acquired brain injury. This gait deviation is characterized by reduced knee flexion during swing phase of the gait cycle and adversely impacts safe foot clearance. Stiff knee gait is an inefficient gait pattern and slows walking speed, limiting one's ability to adapt walking to community mobility demands. Fall risk is increased with this gait problem due to low or ineffective foot clearance. Common compensatory strategies are employed, such as circumduction, hip hiking or vaulting, during ambulation.

The purpose of this study is to examine both the immediate (one month post-injection) and longer-term (4 months post-injection) effects of botulinum toxin injections to the rectus femoris (RF) on gait function in persons with brain injury. This study is clinically important to help inform rehabilitation professionals regarding treatment decisions for management of inefficient and often unsafe stiff knee gait problems following brain injury.

Research Questions:

* Is there a statistically significant difference in mean peak knee flexion between the experimental and control group?
* Is there a statistically significant difference in mean peak knee velocity during the preswing and initial swing phases of gait between the experimental and control group?
* Is there a statistically significant difference in gait function (based on 6-Minute Walk time and temporal distance measures) between the experimental and control group?

DETAILED DESCRIPTION:
Pathophysiologic factors that may contribute to stiff knee gait in persons with brain injury are muscle hypertonicity of the quadriceps muscles, hip flexor weakness, and over activity of the gastrocsoleus muscles in terminal stance(1). Kerrigan et al (2) reported that hyperactivity of the Rectus Femoris (RF) during swing phase was a key contributor to this dynamic swing phase deficit in adults with spastic paresis. Overactivity of the RF muscle during early swing phase has also been identified as a major contributor to stiff knee gait dysfunction in children with cerebral palsy (3). Recognition of the role of RF over-activity in stiff knee gait in the cerebral palsy population has led to surgical and medical interventions aimed to minimize this constraint on swing phase mechanics, such as RF transfers, RF release, and Botulinum toxin injections (BTX-A)(4,5). Research in the cerebral palsy population supports the application of these interventions to improve knee flexion during swing phase and improve overall gait function and efficiency (6).

The applicability of these directed interventions for stiff knee gait, particularly the less invasive BTX-A injections to RF, has not been well examined in adults with spastic paresis. Two research groups (7,8) examined the immediate effects of a motor branch block of RF in persons post-stroke with stiff knee gait and reported improved maximum knee flexion and mean knee flexion velocity during preswing and swing phase following the block. Very few studies9,10 to date examined the short-term effects of BTX-A injection to RF on gait function and energy cost during walking in persons post-stroke who ambulated with stiff knee gait. Stoquart and colleagues9 found that at two months following BTX-A injections, subjects had improved maximum knee flexion during swing phase and improved knee flexion velocity during toe off. Energy cost improved only in that subset of subjects who had greater than 10 degrees of knee flexion during swing phase prior to BTX-A injections. The results of this prospective observational study provided initial support for the efficacy of BTX-A intervention for stiff knee gait in adults post-stroke, however, the authors only examined the short-term effects of this intervention(9). Also, this study had limitations in its methodology, as gait function pre- and post-BOTOX® intervention was assessed using an automated treadmill as opposed to gait analysis during overground walking at self selected gait speed. Further research is needed to determine if there is longer-term benefit of BTX-A injections to RF on gait function in the brain injury population.

Research Design:

* Double-blind randomized controlled trial
* Subjects will be randomly assigned to experimental or control group
* The experimental group will receive BTX-A injection to rectus femoris (RF) followed by usual care
* The control group will receive saline injection to RF followed by usual care
* Subjects and researchers will be blinded to group assignment
* Three-dimensional computerized gait assessments will be conducted pre-treatment (within 2 weeks prior to BOTOX®/placebo injection), 1 month post and 4 months post-injection

ELIGIBILITY:
Inclusion Criteria:

* Greater than 6 months post-acquired brain injury
* Male or female subjects, at least 18 years of age
* Independent ambulation with or without assistive device or orthotic device
* Cognitive Rancho Level VI or higher, ability to follow directions, and likely to complete all required visits
* At least 100 degrees of passive knee flexion ROM
* Gait velocity greater than or equal to 0.4 m/sec
* Modified Ashworth scale rating of 1+ or higher for RF spasticity
* Written informed consent and/or assent has been obtained
* Meet criteria for stiff knee gait based on baseline computerized gait analysis data less than 2 weeks prior to receiving intervention, including:

  * Peak knee flexion less than or equal to 50 degrees (or > 2 standard deviations below normal adult peak knee flexion)
  * Peak knee flexion velocity less than or equal to 256 degrees/% gait cycle (or > 2 standard deviations below normal peak knee flexion velocity)

Exclusion Criteria:

* Change in spasticity medications during course of the study
* Ankle plantarflexion contracture greater than 0 degrees
* Females with a positive pregnancy test, or who are breast-feeding, planning a pregnancy during the study, who think that they may be pregnant at the start of the study or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study
* Has had treatment with botulinum toxin of any serotype to RF or gastrocsoleus up to 12 months prior to enrollment in study
* Evidence of current alcohol or drug abuse or history of neuropsychiatric condition not related to ABI
* Concurrent participation in another investigational drug or device study up to12 months prior to enrollment in study
* Infection or skin disorder at an anticipated injection site
* Uncontrolled clinically significant medical condition other than the condition under evaluation
* Known allergy or sensitivity to any of the components in the study medication, including human serum albumin and sodium chloride as well as the botulinum toxin protein
* Any medical condition that may put the subject at increased risk with exposure to BOTOX including, but not limited to, diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, peripheral neuropathy or any other disorder that might interfere with neuromuscular function
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krisanne B Chapin, PhD, Principal Investigator — Mary Free Bed Rehabilitation Hospital; Cathy Harro, PT, MS, NCS, Principal Investigator — Grand Valley State University
Locations (1):
- Mary Free Bed Rehabilitation Hospital, Grand Rapids, Michigan, United States

REFERENCES:
- [Background] 1. Perry J. Gait Analysis: Normal and Pathological Function. 1st Ed. Thorofare, NJ: SLACK Incorporated; 1992.
- [Background] Kerrigan DC, Gronley J, Perry J. Stiff-legged gait in spastic paresis. A study of quadriceps and hamstrings muscle activity. Am J Phys Med Rehabil. 1991 Dec;70(6):294-300. PMID 1741998
- [Background] Sutherland DH, Davids JR. Common gait abnormalities of the knee in cerebral palsy. Clin Orthop Relat Res. 1993 Mar;(288):139-47. PMID 8458127
- [Background] Perry J. Distal rectus femoris transfer. Dev Med Child Neurol. 1987 Apr;29(2):153-8. doi: 10.1111/j.1469-8749.1987.tb02130.x. PMID 3582785
- [Background] Ward AB, Molenaers G, Colosimo C, Berardelli A. Clinical value of botulinum toxin in neurological indications. Eur J Neurol. 2006 Dec;13 Suppl 4:20-6. doi: 10.1111/j.1468-1331.2006.01650.x. PMID 17112346
- [Background] Cosgrove AP, Corry IS, Graham HK. Botulinum toxin in the management of the lower limb in cerebral palsy. Dev Med Child Neurol. 1994 May;36(5):386-96. doi: 10.1111/j.1469-8749.1994.tb11864.x. PMID 8168657
- [Background] Chantraine F, Detrembleur C, Lejeune TM. Effect of the rectus femoris motor branch block on post-stroke stiff-legged gait. Acta Neurol Belg. 2005 Sep;105(3):171-7. PMID 16255155
- [Background] Sung DH, Bang HJ. Motor branch block of the rectus femoris: its effectiveness in stiff-legged gait in spastic paresis. Arch Phys Med Rehabil. 2000 Jul;81(7):910-5. doi: 10.1053/apmr.2000.5615. PMID 10896003
- [Background] Stoquart GG, Detrembleur C, Palumbo S, Deltombe T, Lejeune TM. Effect of botulinum toxin injection in the rectus femoris on stiff-knee gait in people with stroke: a prospective observational study. Arch Phys Med Rehabil. 2008 Jan;89(1):56-61. doi: 10.1016/j.apmr.2007.08.131. PMID 18164331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting began in January of 2008 and concluded June 1, 2011. Recruiting sites included:inpatient and outpatient settings of a rehabiliation hospital, local support groups, assisted living and retirement homes. Target of N=60 (30 in each arm) was not met.
Pre-assignment Details: Strict inclusion criteria (e.g., walking velocity, rectus femoris spasticity, and target kinematic aspects of peak knee flexion in swing) eliminated many potential participants. 72 participants screened by phone, 30 declined/disqualified, 42 underwent clinical and gait analysis baseline screening, 23 disqualified. A total of 19 were enrolled
Groups:
- Botulinum Toxin Injection to Rectus Femoris: botulinum toxin A (BTX-A) : 200 Units BTX-A reconstituted with 2 cc sterile normal saline in 100:1 ratio. Teflon-coated EMG guidance for confirmation of injection into the Rectus femoris muscle in addition to utilizing standardized injection landmarks, the solution will be injected in 0.5 cc aliquots into 4 different injectate sites within the muscle.
- Saline Injection to Rectus Femoris: placebo : A total of 2 cc sterile normal saline: will be injected in 0.5 cc aliquots into 4 different injectate sites within the rectus femoris (with EMG guidance) of the involved limb.
Period: Overall Study
Arm/Group | Botulinum Toxin Injection to Rectus Femoris | Saline Injection to Rectus Femoris
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Injection to Rectus Femoris | Saline Injection to Rectus Femoris | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 3 | 1 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (17.5) | 49.8 (15.6) | 48.9 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Peak Knee Flexion During Swing Phase of Gait
Description: Measured via computerized gait analysis, the average of peak knee flexion during swing phase.
Time Frame: baseline, 1-month and 4-month post-injection
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Botulinum Toxin Injection to Rectus Femoris | Saline Injection to Rectus Femoris
Number analyzed (Participants) | 10 | 9
degrees
  Peak knee flexion, 1-month post-injection | 31.6 (11.8) | 30.8 (14.3)
  Peak knee flexion, 4-month post-injection | 32.8 (11.0) | 28.5 (14.5)
  Peak knee flexion, Baseline | 29.2 (11.7) | 29.1 (12.4)
Statistical Analysis 1: Comparison: Botulinum Toxin Injection to Rectus Femoris vs Saline Injection to Rectus Femoris; ANOVA; Test type: Non-Inferiority or Equivalence — a priori power calculation suggested N=26 for each group; p = 0.761, ANOVA — p<0.05 threshold; Correlations with walking speed and time since injury were initially performed to determine whether ANCOVA would be be more appropriate

2. Secondary Outcome: Gait Function (Based on 6-Minute Walk)
Description: Average walking speed as calculated during a 6-min walk
Time Frame: baseline, 1-mo and 4-mo post-injection
Population: intention to treat
Measure: Mean (Standard Deviation); unit: meters/sec
Arm/Group | Botulinum Toxin Injection to Rectus Femoris | Saline Injection to Rectus Femoris
Number analyzed (Participants) | 10 | 9
meters/sec
  6min walk test, average speed, baseline | .72 (.18) | .65 (.27)
  6min walk test, average speed, 1M post-inj | .69 (.21) | .70 (.31)
  6min walk test, average speed, 4M post-inj | .69 (.19) | .71 (.26)
Statistical Analysis 1: Comparison: Botulinum Toxin Injection to Rectus Femoris vs Saline Injection to Rectus Femoris; Test type: Superiority or Other; p = .896, ANOVA

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Injection to Rectus Femoris | Saline Injection to Rectus Femoris
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
Early termination due to difficulty identifying and recruiting participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No